CLINICAL TRIAL: NCT05960578
Title: TRAMP: Tumor Necrosis Factor- α Blockade and AR Inhibition in Men With CRPC
Brief Title: Golimumab and Apalutamide for the Treatment of Castration-Resistant Prostate Cancer, TRAMP Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1123487; NCI-2023-04887 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020135 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-Resistant Prostate Carcinoma; Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Biopsy; Specimen Handling; golimumab; Immunoglobulin G; Disulfides; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (golimumab, apalutamide) (Experimental): Patients receive golimumab SC every 4 weeks for 6 doses and apalutamide PO daily. Treatment with apalutamide continues in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy at baseline and during cycle 4. Patients also undergo CT scans or MRI, PSMA PET, bone scan, and collection of blood samples throughout the study.
  Interventions: Drug: Apalutamide; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Golimumab; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Procedure: Bone Scan

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Golimumab — Given SC
  Other Names: CNTO 148; Immunoglobulin G1, Anti-(Human Tumor Necrosis Factor Alpha) (Human Monoclonal CNTO 148 Gamma-1-Chain), Disulfide with Human Monoclonal CNTO 148 Kappa-Chain, Dimer
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: PSMA PET Scan — Undergo PSMA PET
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy

SUMMARY:
This phase II trial tests how well golimumab and apalutamide work in treating patients with castration resistant prostate cancer. Golimumab is in a class of medications called tumor necrosis factor (TNF) inhibitors. It works by blocking the action of TNF, a substance in the body that causes inflammation. Apalutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of cancer cells. Giving golimumab and apalutamide may work better in treating patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive golimumab subcutaneously (SC) every 4 weeks for 6 doses and apalutamide orally (PO) daily. Treatment with apalutamide continues in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy at baseline and during cycle 4. Patients also undergo computed tomography (CT) scans or magnetic resonance imaging (MRI), prostate-specific membrane antigen (PSMA) positron emission tomography (PET), bone scan, and collection of blood samples throughout the study.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically diagnosed prostatic adenocarcinoma
* Participants must have progressed on no more than one novel hormonal therapy (NHT) by PSA or radiographic criteria (per Prostate Cancer Working Group 3 [PCWG3] or Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1) and a castrate serum testosterone level (i.e., ≤ 50 ng/dL). If progressive disease by radiographic criteria, PSA must be ≥ 2ng/ml. PSA progression will be defined as at least two successive PSA rises above the nadir, separated by ≥ 1 week, with the last determination having a value of ≥ 2 ng/mL. NHTs include but are not limited to either abiraterone, enzalutamide, darolutamide, or apalutamide. (Biosimilar or generic agents may be allowed at the discretion of the principal investigator [PI].) Note: prior NHT exposure that did not result in disease progression will not be counted as prior line, i.e., patient's that completed prior abiraterone course in the localized setting, patients that changed NHT due to toxicity or financial toxicity
* Participants must have previously progressed on a novel hormonal therapy (NHT) by PSA or radiographic criteria (per PCWG3 or RECIST v1.1). NHTs include but are not limited to either abiraterone, enzalutamide, darolutamide, or apalutamide. (Biosimilar or generic agents may be allowed at the discretion of the principal investigator [PI].) Note: prior NHT exposure that did not result in disease progression will not be counted as prior line, i.e., patient's that completed prior abiraterone course in the localized setting, patients that changed NHT due to toxicity or financial toxicity
* Participants may have received one prior line of taxane chemotherapy in any setting
* Participants must be >= 18 years of age prior to signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status score =< 2
* Hemoglobin >= 9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
* Platelet count >= 100,000 x 10^9/uL independent of transfusion and/or growth factors within 3 months prior to randomization
* Absolute neutrophil count >= 1.5 x 10^3/mL
* Serum albumin >= 3.0 g/dL
* Serum creatinine =< 1.5 mg/dL
* Serum potassium >= 3.5 mmol/L
* Serum total bilirubin < 1.5 x upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase =< 1.5 x ULN
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug
* Medications known to lower the seizure threshold (see list under prohibited meds) must be discontinued or substituted at least 4 weeks prior to study entry
* Have had no known recent close contact with a person with active tuberculosis (TB) or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation
* Participants must sign an informed consent form (ICF) indicating that they understand the purpose of, and procedures required for, the study and are willing to participate in the study

Exclusion Criteria:

* Subjects may not be receiving other investigational agents within 14 days prior to enrollment
* Subjects with predominant small cell or neuroendocrine variant prostate cancer on most recent standard of care biopsy
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition that could interfere with patient safety
* Symptomatic central nervous system (CNS) metastases. Treated CNS metastases will be allowed if these are stable for at least 8 weeks prior to enrollment
* Uncontrolled or active infection, including:

  * Hepatitis B infection (acute or chronic) as defined according to the American Society of Clinical Oncology guidelines, or hepatitis C infection (anti-hepatitis C virus [HCV] antibody positive and HCV-ribonucleic acid [RNA] quantitation positive)
  * Recent serious infection (e.g., requiring IV antibiotics or hospitalization within last two months)
  * Herpes zoster infection within 2 months of screening
  * History of active granulomatous infection, including histoplasmosis, or coccidioidomycosis
  * HIV (HIV antibody positive)
  * Active or untreated latent tuberculosis
  * History of infected joint prosthesis or received antibiotics for suspected infection of a joint prosthesis in the past five years, if that prosthesis has not been removed or replaced
  * Less serious infections (e.g., acute upper respiratory tract infection, simple urinary tract infection) need not be considered exclusionary at the discretion of the investigator
* Has impaired wound healing capacity defined as current skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions
* Major surgery within 2 weeks of the first dose, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study or within 2 weeks after the last dose of study drug administration (Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate)
* Co-administration of other TNF-alpha inhibitors or disease-modifying anti-rheumatic drugs (DMARDS) for the treatment of rheumatoid arthritis or other rheumatologic condition. (Note: prior exposure to TNF-alpha inhibitors is allowed for non-rheumatologic disease (e.g., SARS-CoV-2) if washout period > 5 half-lives prior to study enrollment)
* Any other issue that would impair the ability of the subject to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Presence of significant cardiovascular disease including New York Heart Association (NYHA) class II-IV heart failure, uncontrolled arrhythmia, myocardial infarction (MI) or stroke within 6 months
* History of autoimmune disorder, including multiple sclerosis or optic neuritis, lupus or lupus-like Syndrome
* Hypersensitivity to any biologics or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies (mAbs), or antibody fragments
* Have a transplanted organ (with the exception of a corneal transplant performed > 3 months prior to first administration of study drug)
* Currently has a malignancy or a history of malignancy within 3 years before screening (with the exception of prostate cancer, treated superficial bladder cancer, or a nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months prior to the administration of the first study intervention
* Immune deficiency syndrome (e.g., severe combined immunodeficiency syndrome [SCIDS], T cell deficiency syndromes, B cell deficiency syndromes, and chronic granulomatous disease)
* Have had a Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening. Patients must agree not to receive BCG vaccination during the study and within 16 weeks after the last administration of study intervention
* Known allergies, hypersensitivity, or intolerance to apalutamide or its excipients
* Gastrointestinal disorder affecting absorption
* History of seizure or any condition that in the opinion of the investigator may predispose to seizure or treatment with drugs known to lower the seizure threshold within 4 weeks prior to starting treatment with apalutamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate specific antigen (PSA)50 response rate | Up to 12 weeks
  Defined by at least a 50% decline in PSA from baseline, in subjects with castrate resistant prostate cancer after combination treatment with TNF-alpha alpha blockade (golimumab) and AR antagonism (apalutamide).

SECONDARY OUTCOMES:
Objective response rate | Up to 4 years
  Will determine objective response rate of measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors version 1.1 criteria for soft tissue metastases.
Radiographic progression free survival (PFS) | Up to 4 years
  The sample mean and standard errors of the time to radiographic progression after the treatment will be summarized, and the post-treatment radiographic response rate together with its 95% confidence interval will be reported.
PSA PFS | Up to 4 years
  The interval between enrollment and the date of documented PSA progression. Progression will be declared if patient has documented to have a testosterone less than 50 ng/dL. In cases where a testosterone level has not been obtained and patient has not had an orchiectomy, progressive disease will be deemed if patient had a documented rise in PSA on luteinizing hormone-releasing hormone analogue therapy. Progression free survival curves will be generated using Kaplan-Meier method.
PSA Doubling Time | Up to 4 years
  The rate of PSA doubling will be calculated from nadir to confirmed PSA progression after 2 subsequent rises 1 week apart using standard calculators
Time to subsequent antineoplastic therapy | Up to 4 years
  The interval between enrollment and the date of documented initiation of next therapy.
Incidence of adverse events | Up to 30 days after final receipt of golimumab administration
  Assess the incidence and severity of adverse events according to the National Cancer Institute - Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Raychaudhuri, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No